CLINICAL TRIAL: NCT05666466
Title: Noninvasive Diagnostic Techniques in Determination of Site of Lesion of Auditory Neuropathy Spectrum Disorder(ANSD)
Brief Title: Noninvasive Diagnostic Techniques in Determination of Site of Lesion of Auditory Neuropathy Spectrum Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Rania Fattouh Ahmad Khalil, Principal investigator, Sohag University
Other Study IDs: Soh-Med-22-12-16
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Auditory Neuropathy
Keywords: auditory neuropathy
MeSH Terms: conditions — Auditory neuropathy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- case group: age between 12 to 50 disproportionate SRS to PTA level presence of OAE presence of CM Normal MRI and CT
  Interventions: Diagnostic Test: extratympanic electrocochleograhy
- control group: age and sex matched to study group Normal hearing sensitivity and excellent speech discrimination no CAPD
  Interventions: Diagnostic Test: extratympanic electrocochleograhy

INTERVENTIONS:
Diagnostic Test: extratympanic electrocochleograhy — electrophysiological test
  Other Names: EchoG

SUMMARY:
cross-sectional study of population who have ANSD

DETAILED DESCRIPTION:
Cross-sectional nonivasive study including study and control group aiming to determine site of lesion of auditory neuropathy spectrum disorder either presynaptic or postsynaptic by using electrophysiological measures

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 50 years OAE and CM could be present disproportionate SRS to PTA level

Exclusion Criteria:

proportionate ABR to PTA level Proportionate SRS to PTA level

* presnce ol lesions in CT or MRI

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 25 participants aged between 12 to 50 years old with disproportionate SRS to PTA level, ABR may be absent or with disturbed waves or wave 5 could be detected at high intense stimulus, OAE and CM could be present. CT and MRI are free
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
determination of site of lesion of ANSD | one and half year
  differentiation between presynaptic and postsynaptic types of ANSD

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag Faculty of Medicine, Sohag, Egypt